CLINICAL TRIAL: NCT03444935
Title: Phone Call Follow-up After Crisis Centre Presentation With Suicidal Ideation and Behaviours.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Winnipeg Regional Health Authority (Other)
Collaborators: Primary Supervisor: Dr. James Bolton MD FRCPC (Unknown)
Responsible Party: Principal Investigator, Laura Sutherland, PGY1 Psychiatry (University of Manitoba), Winnipeg Regional Health Authority
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PCF2018
Record Dates: First submitted 2018-02-19; First posted 2018-02-26 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Suicide; Suicidal Ideation; Suicide, Attempted; Suicide Gesture; Suicide and Self-harm
Keywords: Phone; Brief Contact Intervention; Caring Contact; Follow-up; Suicide; Suicidal Ideation; Suicidal Behaviour; Suicide Attempt
MeSH Terms: conditions — Suicide; Suicidal Ideation; Suicide, Attempted; Self-Injurious Behavior

STUDY DESIGN:
Intervention Model Description: Participants are randomized to one of two groups: intervention or control. Participants will receive a set number of follow-up phone calls based on the group to which they are randomized.
Who Masked: Participant
Masking Description: Crisis Clinicians who consent individuals for participation will be masked from randomization. The randomization process will be completed by a different staff member separate from the Crisis Clinician to prevent allocation bias.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): Participants randomized to the intervention group will receive a predetermined amount of follow-up phone calls after discharge from the Crisis Centre. They can expect a minimum of one call and a maximum of five calls over the five week period immediately following discharge to the community. The number and nature of phone calls they receive will be different from participants in the control group. Participants will be informed upon discharge of the dates they should anticipate phone calls, but it will not be revealed to them which group they were randomized to.
  Interventions: Behavioral: Follow-up phone call
- Control (Other): Participants randomized to the control group will receive a predetermined amount of follow-up phone calls after discharge from the Crisis Centre. They can expect a minimum of one call and a maximum of five calls over the five week period immediately following discharge to the community. The number and nature of phone calls they receive will be different from participants in the intervention group. Participants will be informed upon discharge of the dates they should anticipate phone calls, but it will not be revealed to them which group they were randomized to.
  Interventions: Behavioral: Follow-up phone call

INTERVENTIONS:
Behavioral: Follow-up phone call — Please see arm/group description.

SUMMARY:
This goal of this research is to examine the efficacy and feasibility of starting a phone call follow-up program for individuals discharged to the community after presenting to the Crisis Response Centre (CRC), a standalone mental health facility in Winnipeg, with suicidal ideation or behaviours. Currently there is no worldwide gold standard for how best to follow-up with individuals following presentations to health services with suicidal ideation or behaviours, despite the period immediately after discharge from mental health services being identified as a period of increased risk for death by suicide (Chung et al., 2017; Steeg et al., 2012). This risk is higher still for individuals who specifically had suicidal ideation or behaviours as a component of their reason for presenting to mental health services (Chung et al., 2017). One strategy that has been employed to mitigate this risk is brief contact interventions (BCI), which involves following up with people through text, phone calls, or written messages. Research has shown that this type of follow-up is well-received by individuals and although some studies have found this strategy reduces the rates of suicidal behaviours during this high-risk period, the overall literature shows mixed results (Miller et al., 2017; Exbrayat et al., 2017; Cebria et al., 2016; Milner et al., 2015; Morthorst et al., 2012; Fleischmann et al., 2008; Cedereke et al., 2002).

Because the research on phone call follow up programs has been mixed, we will be conducting a brief trial to study the efficacy and feasibility of a phone call follow-up system in Winnipeg to inform whether or not this type of program would be of benefit to the community. In order to best study this, we will be conducting a randomized control trial for individuals who are discharged to the community after presenting to the CRC with a recent history of suicidal thoughts or behaviours. Participants will be randomized into either an intervention group or a control group. All participants will receive at least one and no more than five phone calls during the five-week period immediately following discharge from the CRC, and the content and timing of these phone calls will be different depending on which group a participant is randomized to. We will rely on both self-reported data, which will be collected in a formalized fashion, and data in the electronic medical records of participants to analyze this intervention. Our hypothesis is that the specific protocol we have designed to follow up with the intervention group will result in decreased suicidal thoughts and behaviours in the period immediately following discharge.

DETAILED DESCRIPTION:
The proposed randomized control trial will occur over a three-month period at the Crisis Response Centre (CRC) in Winnipeg. The CRC serves as a standalone facility that offers 24/7 walk in assessment and treatment for adults with mental health crises, as well as referrals to mental health services. All individuals who present to the CRC and report any suicidal ideation or behaviour within the one week prior to their presentation will be considered eligible for the study. Further inclusion and exclusion criteria are outlined in the "Eligibility" section. A variety of employees at the CRC will be involved in different roles to assist with this research.

In current practice, all individuals are able to connect with Crisis Clinicians working at the CRC both in person and through the use of a telephone call to the Mobile Crisis Unit, which provides the capacity for Crisis Clinicians to both talk on the phone to individuals or leave the CRC and assess individuals offsite to support them. All individuals who connect with Crisis Clinicians in any of these capacities have a Mental Health Assessment (MHA) completed by Crisis Clinicians. All Crisis Clinicians are trained specifically in how to assess and assist individuals with suicidal thoughts or behaviours, therefore making them optimal individuals to assist in this research given their experience to support the safety of individuals in crisis.

Participants who present to the CRC, are deemed appropriate for participation in the study based on inclusion and exclusion criteria, and who are otherwise ready for discharge back into the community will be consented by the same Crisis Clinician who completed their MHA. Participants will be informed that they will receive no less than one and no more than five phone calls over the five weeks immediately following the date of their discharge from the CRC as part of this study, without informing them of the specific differences between the intervention and control groups. Individuals will decide prior to discharge whether they would like to participate, and those who choose to participate will provide a phone number that they can be contacted at and that messages can be left on.

Individuals who choose to participate will be randomized to either a control or intervention group based on a coin flip done by the Attendants (Front Desk Staff at the CRC). The Crisis Clinician will not be involved in the randomization process to prevent allocation bias. Once participants are randomized, they will be informed by the Attendants of the exact dates on which they should expect phone calls without revealing to the participant what group they have been randomized to, thereby blinding the participants. This blinding is possible because we have concealed the exact number and nature of phone calls that will occur for the two groups. Attendants will update a schedule after randomizing each participant with appointment times for all phone calls required for the study.

On each day, Team Leads will be responsible for reviewing the schedule and allocating all required phone calls between themselves and the Crisis Clinicians working that day. Crisis Clinicians will attempt to call participants a maximum of three times on the assigned day between 0800 and 2200. All Crisis Clinicians are provided with scripts to follow for phone calls based on which group they are calling and at what time. If Crisis Clinicians are unsuccessful at contacting the participant by the third attempt, they will leave a scripted voicemail offering support and encouraging the participant to call back. If at any point during phone conversations the Crisis Clinician has concerns about a participant's safety or suicide risk, this will be approached in the same way the Clinician would approach anyone who calls in to the Mobile Crisis Unit with suicidal ideation or behaviours.

Crisis Clinicians will record the outcome and content of all phone calls into the electronic medical record, including phone calls where they do and do not successfully talk with the participant. Throughout the study, Dr. Laura Sutherland will be reviewing the participants' electronic medical records with particular attention to mental health diagnoses, visit history during the study time, and the notes from all phone calls made. This information will be used to analyze all of the data in a deidentified fashion. Crisis Clinicians and Team Leads will also keep a daily tally of the total number of individuals considered appropriate for the study based on inclusion and exclusion criteria, and how many of these individuals decline participation in the study to further inform the analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Being discharged to the community from the Crisis Centre
2. At least 18 years old
3. Suicidal ideation or behaviour within one week of presentation to the CRC

   1. Suicidal ideation = thoughts of suicide or death, ranging from passive thoughts to organized plans
   2. Suicidal behaviour = suicide attempt, interrupted suicide attempt, aborted suicide attempt, suicide preparatory actions (eg. writing a suicide note, selling off/giving away all possessions)

Exclusion Criteria:

1. Medically or cognitively unable to participate
2. Having an insurmountable language barrier
3. Psychiatrist deems that this type of follow-up could be harmful for the patient
4. Living in an institutional setting
5. Patient being admitted to hospital/treatment facility as a result of their presentation to the Crisis Response Centre
6. Being enrolled in outreach/follow up program that would directly overlap with involvement in this study
7. No reliable access to phone

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2018-05-14 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2025-03-20 (Actual)

PRIMARY OUTCOMES:
Suicidal ideation (frequency) | Self-report; outcome pertains to frequency over the entire five weeks.
  Self-report of any thoughts of ending own life, from passive thoughts to formal plans.
Suicidal behaviours (frequency) | Self-report; outcome pertains to frequency over the entire five weeks.
  Self-report that includes a gradation of behaviour: suicide attempt, interrupted attempt, aborted attempt, or suicide preparatory act (eg. writing suicide note, selling off possessions). Note that death by suicide is also included in this category (but will only be available if family/friends of participant reports).

SECONDARY OUTCOMES:
Non-suicidal self harm (frequency) | Self-report; outcome pertains to frequency over the entire five weeks.
  Self-report of any self-harm without the intention of ending own life.
Health care utilization (frequency) | Self-report; outcome pertains to frequency over the entire five weeks.
  Self-report of any health care utilization, including Crisis Centre, Emergency Department, Urgent Care, Crisis Hotlines, Family Physician, Walk In Clinics. Also collected through review of visit history with entrance complaint in electronic medical records.
Perceived mental health | Self-report; outcome pertains to frequency over the entire five weeks.
  Self-report of mental health using Likert-scale questioning
Perceived improvement in mental health | Self-report; outcome pertains to perceived improvement since the date of enrollment.
  Self-report of perceived improvement in mental health using Likert-scale questioning
Satisfaction with and perceived helpfulness of phone calls in reducing suicidal thoughts and behaviours. | Self-report; outcome pertains to frequency over the entire five weeks.
  Self-report of satisfaction with, perceived helpfulness of phone call follow-ups in reducing suicidal thoughts and behaviours using Likert-scale questions

CONTACTS AND LOCATIONS:
Overall Officials: Laura Sutherland, MD, Principal Investigator — Winnipeg Regional Health Authority
Locations (1):
- Crisis Response Centre, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chung DT, Ryan CJ, Hadzi-Pavlovic D, Singh SP, Stanton C, Large MM. Suicide Rates After Discharge From Psychiatric Facilities: A Systematic Review and Meta-analysis. JAMA Psychiatry. 2017 Jul 1;74(7):694-702. doi: 10.1001/jamapsychiatry.2017.1044. PMID 28564699
- [Background] Steeg S, Kapur N, Webb R, Applegate E, Stewart SL, Hawton K, Bergen H, Waters K, Cooper J. The development of a population-level clinical screening tool for self-harm repetition and suicide: the ReACT Self-Harm Rule. Psychol Med. 2012 Nov;42(11):2383-94. doi: 10.1017/S0033291712000347. Epub 2012 Mar 7. PMID 22394511
- [Background] Fleischmann A, Bertolote JM, Wasserman D, De Leo D, Bolhari J, Botega NJ, De Silva D, Phillips M, Vijayakumar L, Varnik A, Schlebusch L, Thanh HT. Effectiveness of brief intervention and contact for suicide attempters: a randomized controlled trial in five countries. Bull World Health Organ. 2008 Sep;86(9):703-9. doi: 10.2471/blt.07.046995. PMID 18797646
- [Background] Milner AJ, Carter G, Pirkis J, Robinson J, Spittal MJ. Letters, green cards, telephone calls and postcards: systematic and meta-analytic review of brief contact interventions for reducing self-harm, suicide attempts and suicide. Br J Psychiatry. 2015 Mar;206(3):184-90. doi: 10.1192/bjp.bp.114.147819. PMID 25733570
- [Background] Miller IW, Camargo CA Jr, Arias SA, Sullivan AF, Allen MH, Goldstein AB, Manton AP, Espinola JA, Jones R, Hasegawa K, Boudreaux ED; ED-SAFE Investigators. Suicide Prevention in an Emergency Department Population: The ED-SAFE Study. JAMA Psychiatry. 2017 Jun 1;74(6):563-570. doi: 10.1001/jamapsychiatry.2017.0678. PMID 28456130
- [Background] Cebria AI, Parra I, Pamias M, Escayola A, Garcia-Pares G, Punti J, Laredo A, Valles V, Cavero M, Oliva JC, Hegerl U, Perez-Sola V, Palao DJ. Effectiveness of a telephone management programme for patients discharged from an emergency department after a suicide attempt: controlled study in a Spanish population. J Affect Disord. 2013 May;147(1-3):269-76. doi: 10.1016/j.jad.2012.11.016. Epub 2012 Dec 6. PMID 23219058
- [Background] Exbrayat S, Coudrot C, Gourdon X, Gay A, Sevos J, Pellet J, Trombert-Paviot B, Massoubre C. Effect of telephone follow-up on repeated suicide attempt in patients discharged from an emergency psychiatry department: a controlled study. BMC Psychiatry. 2017 Mar 20;17(1):96. doi: 10.1186/s12888-017-1258-6. PMID 28320345
- [Background] Morthorst B, Krogh J, Erlangsen A, Alberdi F, Nordentoft M. Effect of assertive outreach after suicide attempt in the AID (assertive intervention for deliberate self harm) trial: randomised controlled trial. BMJ. 2012 Aug 22;345:e4972. doi: 10.1136/bmj.e4972. PMID 22915730
- [Background] Cedereke M, Monti K, Ojehagen A. Telephone contact with patients in the year after a suicide attempt: does it affect treatment attendance and outcome? A randomised controlled study. Eur Psychiatry. 2002 Apr;17(2):82-91. doi: 10.1016/s0924-9338(02)00632-6. PMID 11973116